CLINICAL TRIAL: NCT01220466
Title: A Prospective Study to Evaluate the Performance and Acceptability of the iDesign Advanced WaveScan Study(tm) System
Brief Title: Performance and Acceptability of iDesign
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR-108-IDSN
Record Dates: First submitted 2010-09-24; First posted 2010-10-14 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Refractive Error (Experimental)
  Interventions: Device: STAR S4IR LASIK with iDesign Aberrometer

INTERVENTIONS:
Device: STAR S4IR LASIK with iDesign Aberrometer — CustomVue LASIK targeted for emmetropia
  Other Names: CustomVue

SUMMARY:
The results of this trial will demonstrate that the iDesign System performs as intended and is acceptable in a clinical setting.

DETAILED DESCRIPTION:
LASIK treatment across the range of myopia with or without astigmatism, hyperopia with or without astigmatism, and mixed astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any race, and at least 18 years old at the time the consent form is signed.
* The refractive error, based on manifest refraction (adjusted for optical infinity), must be MRSE up to -15.00 D with manifest cylinder between 0.00 and -6.00 D; MRSE up to +9.00 D with cylinder between 0.00 and +6.00 D; or manifest cylinder (from 1.00 to 6.00 D) greater than the magnitude of sphere, and the cylinder and sphere have opposite signs.
* BSCVA of 20/20 or better.
* UCVA:

  * Myopes must be 20/40 or worse.
  * Subjects with Hyperopia or mixed astigmatism, treatment may be based on difficulty maintaining UCVA of 20/40 evidenced by spectacle/contact lens dependence for distance, as documented by the investigator.
* Wavefront diameter ≥ 4.0 mm.
* Sufficient agreement between manifest refraction (adjusted for optical infinity) and iDesign System refraction (sphere, cylinder, and axis) to allow treatment selection and generation of an ablation profile as determined by the investigational iDesign System software.
* Manifest refraction sphere within ± 0.75 D of cycloplegic refraction sphere.
* Anticipated post-operative stromal bed thickness of at least 250 microns, based on pre-operative central corneal pachymetry minus the maximum treatment depth to be ablated (as calculated by the iDesign System) and the intended flap thickness.
* Anticipated post-operative keratometry value (based on pre-operative iDesign System refraction and keratometry) that is appropriate.
* A stable refractive error (based on a previous exam, medical records, or prescription) as compared to the unadjusted pre-operative manifest refraction.
* Subjects who currently wear contact lenses must demonstrate refractive stability in the operative eye. Rigid or toric lenses must be removed for at least 2 weeks and SCL for at least 3 days prior to the first refraction used to establish stability. A second refraction with a change of no more than ± 0.50 D MRSE at least 7 days after baseline.
* Willing and capable of returning for follow-up examinations for the duration of the study.

Exclusion Criteria:

* Women who are pregnant, breast-feeding, or intend to become pregnant over the course of the study, as determined by verbal inquiry, or another condition associated with the fluctuation of hormones that could lead to refractive changes.
* Subjects with an ametropic or amblyopic fellow eye not meeting all inclusion criteria that does not fall within the indications for treatment using the VISX® STAR S4 IR™ Excimer Laser.
* Concurrent use of systemic (including inhaled) medications that may impair healing, including but not limited to: steroids, antimetabolites, isotretinoin (Accutane™) within 6 months of treatment, and amiodarone hydrochloride (Cordarone™) within 12 months of treatment.
* Acute or chronic disease, illness, or treatment that would increase the operative risk (e.g., immuno-compromised, autoimmune disease, connective tissue disease, clinically significant atopic disease, diabetes, etc.).
* Subjects with a cardiac pacemaker, implanted defibrillator, implanted neurostimulator, or any active electrical implants.
* Ocular condition (other than high myopia) that may predispose the subject to future complications, such as history or evidence of active or inactive corneal disease
* Previous intraocular or corneal surgery that might confound the outcome of the study or increase risk to the subject.
* Known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course.
* Concurrent participation in any other clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Tarantino, OD, Study Director — Abbott Medical Optics
Locations (4):
- Canada (4):
  - Clearly LASIK, Victoria, British Columbia
  - Image Plus Laser Eye Center, Winnipeg, Manitoba
  - University of Ottawa Eye Institute, The Ottawa Hospital, Ottawa, Ontario
  - Yonge-Eglington Laser, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One or both eyes of 77 subjects (143 eyes) were treated. This includes a predominance of Caucasian participants and a mean age of 37.2 years.
Groups:
- Hyperopia With or Without Astigmatism: Hyperopia with and without astigmatism with MRSE up to
  +9.00 D, with cylinder between 0.00 and +6.00 D.
- Myopia With or Without Astigmatism: Myopia with and without astigmatism with MRSE up to -15.0D, with cylinder between 0.00 and -6.00 D.
- Mixed Astigmatism: Mixed Astigmatism when the magnitude of cylinder (from 1.0 to 6.0D ) is greater than the magnitude of sphere, and the cylinder and sphere have opposite signs.
Period: Overall Study
Arm/Group | Hyperopia With or Without Astigmatism | Myopia With or Without Astigmatism | Mixed Astigmatism
Started | 11 (19 eyes) | 56 (108 eyes) | 10 (16 eyes)
Completed | 11 (19 eyes) | 56 (108 eyes) | 10 (16 eyes)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperopia With or Without Astigmatism | Myopia With or Without Astigmatism | Mixed Astigmatism | Total
Number analyzed (Participants) | 11 | 56 | 10 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 56 | 10 | 77
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 28 | 4 | 38
  Male | 5 | 28 | 6 | 39
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 56 | 10 | 77

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Uncorrected Visual Acuity (UCVA) of 20/40 or Better.
Time Frame: 6 months
Population: UCVA is reported as percentage of eyes not percentage of subjects achieving UCVA of 20/40 or better
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Myopia With and Without Astigmatism: Myopia with and without astigmatism with MRSE up to -15.0 D, with cylinder between 0.00 and -6.00 D.
- Hyperopia With and Without Astigmatism: Hyperopia with and without astigmatism with MRSE up to +9.00 D, with cylinder between 0.00 and +6.00 D
- Mixed Astigmatism: Mixed Astigmatism when the magnitude of cylinder (from 1.0 to 6.0D) is greater than the magnitude of sphere, and the cylinder and sphere have opposite signs.
Arm/Group | Myopia With and Without Astigmatism | Hyperopia With and Without Astigmatism | Mixed Astigmatism
Number analyzed (Participants) | 56 | 11 | 10
Number analyzed (eyes) | 108 | 19 | 16
percentage of eyes | 100 [97.3 to 100] | 100 [85.4 to 100] | 100 [82.9 to 100]

2. Other Pre Specified Outcome: Percentage of Eyes With Manifest Refraction Spherical Equivalent Within 1.0 D
Time Frame: 6 months
Population: Percent of eyes that achieved manifest refraction spherical equivalent within 1.0 D
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Myopia With and Without Astigmatism | Hyperopia With and Without Astigmatism | Mixed Astigmatism
Number analyzed (Participants) | 56 | 11 | 10
Number analyzed (eyes) | 108 | 19 | 16
percentage of eyes | 99.1 [94.9 to 100] | 89.5 [66.9 to 98.7] | 93.8 [69.8 to 99.8]

3. Other Pre Specified Outcome: Percentage of Eyes With Loss of More Than 2 Lines Best Spectacle Corrected Visual Acuity (BSCVA)
Time Frame: 6 Months
Population: Percent of eyes that lost more than 2 lines of BSCVA.
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Myopia With and Without Astigmatism | Hyperopia With and Without Astigmatism | Mixed Astigmatism
Number analyzed (Participants) | 56 | 11 | 10
Number analyzed (eyes) | 108 | 19 | 16
percentage of eyes | 0 [NA to NA] — Confidence intervals were not calculated because 0% of eyes lost more than 2 lines of BSCVA. | 5.3 [0.1 to 26] | 0 [NA to NA] — Confidence intervals were not calculated because 0% of eyes lost more than 2 lines of BSCVA.

4. Other Pre Specified Outcome: Percentage of Eyes With Best Spectacle Corrected Visual Acuity (BSCVA) Worse Than 20/40
Time Frame: 6 Months
Population: Percentage of eyes with BSCVA worse than 20/40
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Myopia With and Without Astigmatism | Hyperopia With and Without Astigmatism | Mixed Astigmatism
Number analyzed (Participants) | 56 | 11 | 10
Number analyzed (eyes) | 108 | 19 | 16
percentage of eyes | 0 [NA to NA] — Confidence intervals were not calculated because 0% of eyes had BSCVA worse than 20/40. | 0 [NA to NA] — Confidence intervals were not calculated because 0% of eyes had BSCVA worse than 20/40. | 0 [NA to NA] — Confidence intervals were not calculated because 0% of eyes had BSCVA worse than 20/40.

5. Other Pre Specified Outcome: Percentage of Eyes With Induced Manifest Refractive Astigmatism Greater Than 2.00 D of Absolute Cylinder as Compared to the Preoperative Refraction
Description: Induced Manifest Refractive Astigmatism is an increase of astigmatism (cylinder) postoperatively that could be caused by the refractive treatment. An increase of greater than 2.0 D is considered a safety endpoint per ANSI Z80.11-2007.
Time Frame: 6 Months
Population: Percentage of eyes with induced manifest refractive astigmatism greater than 2.00 D of absolute cylinder power
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Myopia With and Without Astigmatism | Hyperopia With and Without Astigmatism | Mixed Astigmatism
Number analyzed (Participants) | 56 | 11 | 10
Number analyzed (eyes) | 108 | 19 | 16
percentage of eyes | 0 [NA to NA] — Confidence intervals were not calculated because 0% of eyes had induced manifest refractive astigmatism greater than 2.00 D of absolute cylinder power. | 0 [NA to NA] — Confidence intervals were not calculated because 0% of eyes had induced manifest refractive astigmatism greater than 2.00 D of absolute cylinder power. | 0 [NA to NA] — Confidence intervals were not calculated because 0% of eyes had induced manifest refractive astigmatism greater than 2.00 D of absolute cylinder power.

ADVERSE EVENTS:
Arm/Group | Hyperopia With and Without Astigmatism | Myopia With and Without Astigmatism | Mixed Astigmatism
Serious Adverse Events (participants affected / at risk) | 1/11 | 2/56 | 0/10
Other Adverse Events (participants affected / at risk) | 2/11 | 4/56 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperopia With and Without Astigmatism (N=11) | Myopia With and Without Astigmatism (N=56) | Mixed Astigmatism (N=10)
Decrease in BSCVA of greater than or equal to two lines (Eye disorders) | 1 (1) | 2 (2) | 0 (0) — Loss of greater than two lines of BSCVA is a SAE in the context of this study. Decrease in BSCVA of greater than or equal to 2 lines (10 letters) not due to irregular astigmatism as shown by hard contact lens refraction, at 3 months or later.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperopia With and Without Astigmatism (N=11) | Myopia With and Without Astigmatism (N=56) | Mixed Astigmatism (N=10)
Corneal epithelial defect (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — Corneal epithelial defect of any kind, involving the keratometry at 1 month or later
Foreign body in the eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Miscreated flap (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
retinal tear/hole (Eye disorders) | 0 (0) | 1 (2) | 0 (0) — One subject in the myopia cohort had a retinal tear/hole in both the right and left eye.
Other - car accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Other - concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other